CLINICAL TRIAL: NCT03050879
Title: Prospective Randomized Controlled Trials on Clinical Outcomes of Indocyanine Green Tracer Using in Laparoscopic Gastrectomy With Lymph Node Dissection for Gastric Cancer
Brief Title: Indocyanine Green Tracer Using in Laparoscopic Gastrectomy With Lymph Node Dissection
Acronym: ICGTinLG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Clinical Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-012
Record Dates: First submitted 2017-01-13; First posted 2017-02-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Stomach Neoplasms; Indocyanine Green
Keywords: Stomach Neoplasms; Indocyanine Green Tracer; Laparoscopic Gastrectomy; Lymph Node Dissection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indocyanine Green Tracer (Experimental): Indocyanine Green Tracer will be used in laparoscopic gastrectomy with lymph node dissection for gastric adenocarcinoma in this group.
  Interventions: Drug: Indocyanine Green Tracer
- No Indocyanine Green Tracer (Active Comparator): Indocyanine Green Tracer will not be used in laparoscopic gastrectomy with lymph node dissection for gastric adenocarcinoma in this group.
  Interventions: Drug: Indocyanine Green Tracer

INTERVENTIONS:
Drug: Indocyanine Green Tracer — Laparoscopic gastrectomy with lymph node dissection for gastric cancer using Indocyanine Green Tracer
  Other Names: ICG

SUMMARY:
The purpose of this study is to explore the clinical outcomes of Indocyanine Green Tracer using in laparoscopic gastrectomy with lymph node dissection for gastric adenocarcinoma（cT1-4a, N-/+, M0）.

DETAILED DESCRIPTION:
Indocyanine Green Tracer is often applied in surgery for early gastric adenocarcinoma. Its application in laparoscopic gastrectomy with lymph node dissection for gastric adenocarcinoma is at the stage of cases accumulation, method studying and clinical research. There is no prospective studies to identify the clinical outcomes of Indocyanine Green Tracer using in laparoscopic gastrectomy with lymph node dissection for gastric adenocarcinoma.

On the basis of more than 3000 cases of laparoscopic gastrectomy with lymph node dissection for gastric adenocarcinoma, we want to apply the Indocyanine Green Tracer, a cheap, easy to operate and no radiation pollution way, to predict the positive lymph nodes in gastric adenocarcinoma, to guid the scope of laparoscopic lymph node dissection for gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* clinical stage tumor 1-4a (cT1-4a), N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values
* Diffuse; widespread; plastica

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-07-13 (Actual); Study Completion 2019-07-13 (Actual)

PRIMARY OUTCOMES:
Total Number of Retrieved Lymph Nodes | 14 days
  Compare total number of retrieved lymph nodes in both group.

SECONDARY OUTCOMES:
The rate of fluorescence | 14 days
  The number of fluorescent lymph node in experimental group is divided by the total number of lymph nodes in active experimental group
Positive rate | 14 days
  The number of positive lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in experimental group
False positive rate | 14 days
  The number of negative lymph nodes in fluorescent lymph nodes is divided by the number of total fluorescent lymph nodes in experimental group
Negative rate | 14 days
  The number of negative lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in experimental group
False negative rate | 14 days
  The number of positive lymph nodes in not fluorescent lymph nodes is divided by the number of total not fluorescent lymph nodes in experimental group
Number of Metastasis Lymph Nodes | 14 days
  Compare number of positive lymph nodes in both group.
Metastasis rate of lymph node | 14 days
  Compare metastasis rate of lymph node in both group
Morbidity and mortality rates | 30 days
  This is for the early postoperative complication and mortality, which defined as the event observed within 30 days after surgery.
3-year disease free survival rate | 36 months
  disease-free survival was defined as the time from surgery to the time of recurrence or death from any cause
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Postoperative recovery course | 10 days
  Time to first ambulation, flatus, liquid diet and soft diet, duration of postoperative hospital stay and postoperative pain are used to assess the postoperative recovery course.Visual analog pain score method is used to evaluate the difference of postoperative pain degree.
Operation time | 1 day
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
Intraoperative blood loss | 1 day
Conversive rate | 1 day
Intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
Incision length | 1 day
The variation of cholesterol | 3, 6, 9 and 12 months
  The variation of cholesterol in millimole/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of album | 3, 6, 9 and 12 months
  The variation of album in gram/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The results of endoscopy | 3, 6, 9 and 12 months
  The incidence of reflux esophagitis under the endoscopy on postoperative 3 and 12 months are used to access the postoperative quality of life.
The variation of body temperature | 8 days
  The daily highest body temperature in degree centigrade before discharge are recorded to access the inflammatory and immune response.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of prealbumin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of prealbumin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
3-year overall survival rate | 36 months
  Overall survival was defined as the time from surgery to death from any cause
5-year overall survival rate | 60 months
  Overall survival was defined as the time from surgery to death from any cause
5-year disease free survival rate | 60 months
  disease-free survival was defined as the time from surgery to the time of recurrence or death from any cause
5-year recurrence pattern | 60 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhong Q, Wu D, Liu ZY, Shang-Guan ZX, Huang ZN, Zhang ZQ, Qiu TY, Chen JY, Jiang YM, Lin GT, Tang YH, Li P, Xie JW, Lin JX, Zheng CH, Chen QY, Huang CM. Long-term oncological outcomes of indocyanine green fluorescence imaging-guided laparoscopic lymphadenectomy for gastric cancer: 5-year outcomes from the FUGES-012 randomized clinical trial. BMC Med. 2025 Aug 26;23(1):497. doi: 10.1186/s12916-025-04334-1. PMID 40859341
- [Derived] Chen QY, Zhong Q, Liu ZY, Li P, Lin GT, Zheng QL, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Zeng GR, Jiang MC, Wang HG, Huang XB, Xu KX, Li YF, Zheng CH, Xie JW, Huang CM. Indocyanine green fluorescence imaging-guided versus conventional laparoscopic lymphadenectomy for gastric cancer: long-term outcomes of a phase 3 randomised clinical trial. Nat Commun. 2023 Nov 16;14(1):7413. doi: 10.1038/s41467-023-42712-6. PMID 37973806
- [Derived] Huang ZN, He QC, Qiu WW, Wu J, Zheng CY, Lin GS, Li P, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Zheng CH, Chen QY, Huang CM, Xie JW. OSATS scoring confirms ICG enhancement of performance in laparoscopic radical gastrectomy: a post-hoc analysis of a randomized controlled trial. Int J Surg. 2024 Jan 1;110(1):342-352. doi: 10.1097/JS9.0000000000000830. PMID 37939147
- [Derived] Chen QY, Xie JW, Zhong Q, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Zheng HL, Li P, Zheng CH, Huang CM. Safety and Efficacy of Indocyanine Green Tracer-Guided Lymph Node Dissection During Laparoscopic Radical Gastrectomy in Patients With Gastric Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):300-311. doi: 10.1001/jamasurg.2019.6033. PMID 32101269